CLINICAL TRIAL: NCT02200939
Title: Post-Market Evaluation of the Rotation Medical Rotator Cuff System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014.05.12
Record Dates: First submitted 2014-07-23; First posted 2014-07-25 (Estimated); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Partial Thickness Supraspinatus Tendon Tear; Full Thickness Supraspinatus Tendon Tear
MeSH Terms: interventions — Sutureless Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Partial-Thickness Tear (Experimental): Intermediate or High partial-thickness tear (PTT) or very small full-thickness tear of the supraspinatus tendon surgically treated by implantation of the bioinductive implant.
  Interventions: Device: Bioinductive implant
- Full Thickness Tear (Experimental): Medium or large full thickness tear (FTT) of the supraspinatus tendon surgically treated with the bioinductive implant adjunctive to surgical repair.
  Interventions: Device: Bioinductive implant; Device: Surgical repair

INTERVENTIONS:
Device: Bioinductive implant
  Other Names: Rotation Medical Rotator Cuff System™; REGENETEN™ Bioinductive Implant System.
Device: Surgical repair — Surgical repair with commercially-available sutures/suture anchors.
  Arms: Full Thickness Tear

SUMMARY:
The purpose of this study is to evaluate bioinduction of new tissue and tendon healing after implantation of the Rotation Medical Bioinductive Implant used as either a standalone device or adjunct to surgical repair in the treatment of supraspinatus tendon tears.

ELIGIBILITY:
INCLUSION CRITERIA

Subjects enrolled in the study MUST meet all of the following criteria:

1. At least 21 years of age
2. Rotator cuff tear requiring surgery that meets either criterion A or B:

   A. Medium or large partial-thickness tear or very small full-thickness tear of the supraspinatus tendon planned for standalone treatment (no surgical repair with sutures/suture anchors) with the bioinductive implant B. Medium or large full-thickness tear primarily of the supraspinatus tendon planned for treatment with the bioinductive implant adjunctive to surgical repair
3. Chronic shoulder pain lasting longer than 3 months unresponsive to conservative therapy including, but not limited to, pain medication, physical therapy and injections
4. MRI of the shoulder within 60 days prior to the study procedure
5. Willing to comply with the prescribed post-operative rehabilitation program
6. Willing to be available for each protocol-required follow-up examination
7. Able to understand the informed consent process, including regulatory requirements such as HIPAA authorization, and document informed consent prior to completion of any study-related procedures
8. Ability to read, understand, and complete subject-reported outcomes in English

EXCLUSION CRITERIA

Subjects enrolled in the study MUST NOT meet any of the following criteria:

1. Massive rotator cuff tears (≥ 5 cm)
2. Acute rotator cuff tears less than 12 months from injury
3. Previous rotator cuff surgery on the index shoulder
4. Instability of the index shoulder
5. Chondromalacia of index shoulder ≥ Grade 3
6. Fatty infiltration of the index shoulder rotator cuff muscle ≥ Grade 2
7. Calcification of the index shoulder rotator cuff
8. Genetic collagen disease
9. History of insulin dependent diabetes
10. History of auto-immune or immunodeficiency disorders
11. History of chronic inflammatory disorders
12. Oral steroid use in last 2 months or injectable steroid use in last 4 weeks
13. History of heavy smoking (> 1 pack per day) within last 6 months
14. Hypersensitivity to bovine-derived materials
15. Females of child-bearing potential who are pregnant or plan to become pregnant during the course of the study
16. Currently involved in any injury litigation or worker's compensation claims relating to the index shoulder
17. Enrolled, or plans to enroll, in another clinical trial during this study that would affect the outcomes of this study
18. History of non-compliance with medical treatment, physical therapy/rehabilitation, or clinical study participation
19. History of cognitive or mental health status that interferes with study participation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2014-08-20 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura England, Study Chair — Smith & Nephew, Inc.
Locations (15):
- United States (15):
  - Southern California Orthopedic Institute, Van Nuys, California
  - Steadman Hawkins Clinic-Denver, Denver, Colorado
  - Holy Cross Hospital Orthopedic Research Institute, Fort Lauderdale, Florida
  - Harbin Clinic Orthopaedics & Sports Medicine Rome, Rome, Georgia
  - OrthoIllinois, LTD, Rockford, Illinois
  - University of Iowa Sports Medicine, Iowa City, Iowa
  - Towson Orthopaedic Associates / University of Maryland St Joseph Med Ctr, Towson, Maryland
  - Great Lakes Orthopaedic Center, Traverse City, Michigan
  - Twin Cities Orthopedics, Edina, Minnesota
  - Princeton Orthopaedic Associates, P.A., Princeton, New Jersey
  - OrthoCarolina Research Institute, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Texas Orthopedic Specialists, P.L.L.C., Bedford, Texas
  - Bone & Joint Clinic of Houston, Houston, Texas
  - ProOrtho Orthopedic Clinic, Kirkland, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started on 20 August 2014 and the study concluded on 24 November 2020 across 15 participating medical clinics in the United States.
Groups:
- Partial-Thickness Tear: Intermediate or High partial-thickness tear (PTT) or very small full-thickness tear (FTT) of the supraspinatus tendon surgically treated by implantation of the bioinductive implant.
Period: Overall Study
Arm/Group | Partial-Thickness Tear | Full Thickness Tear
Started | 33 | 115
Completed | 31 | 104
Not Completed | 2 | 11
Not completed — Participant withdrew consent | 0 | 1
Not completed — Lost to Follow-up | 2 | 9
Not completed — Subject moved out of town and unable to make it back to study | 0 | 1

BASELINE CHARACTERISTICS:
Population: Number of participants after implantation of the REGENETEN Bioinductive Implant for partial-thickness tear (PTT) or full-thickness tear (FTT) that provided data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Partial-Thickness Tear | Full Thickness Tear | Total
Number analyzed (Participants) | 33 | 115 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.60 (10.13) | 60.40 (8.01) | 59.10 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 39 | 53
  Male | 19 | 76 | 95
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Caucasian | 33 | 100 | 133
  Ethnicity: Asian | 0 | 1 | 1
  Ethnicity: Hispanic | 0 | 5 | 5
  Ethnicity: African American | 0 | 9 | 9
Region of Enrollment [Number; unit: participants]
  United States | 33 | 115 | 148
Hand Dominance [Count of Participants; unit: Participants]
  Right | 29 | 103 | 132
  Left | 4 | 12 | 16
Affected Shoulder [Count of Participants; unit: Participants]
  Right | 17 | 78 | 95
  Left | 16 | 37 | 53
Smoking Habit [Count of Participants; unit: Participants]
  Never Smoked | 20 | 81 | 101
  Former Smoker | 12 | 31 | 43
  Current Smoker | 1 | 3 | 4
Employment Status [Count of Participants; unit: Participants]
  Currently employed (working for pay) | 22 | 83 | 105
  Currently unemployed (not working for pay) | 11 | 32 | 43
Tear Size: Partial-Thickness ONLY [Count of Participants; unit: Participants] — Partial-Thickness Tear Size classified using Ellman grading as:
  * Grade 1: Low (less than 3 millimeters deep)
  * Grade 2: Intermediate (3-6 millimeters deep)
  * Grade 3: High (greater than 6 millimeters deep).
  Tear Size for Partial-Thickness Tears assessed by magnetic resonance imaging (MRI). Population: Full Thickness Tear not measured using this classification (i.e. measure applies to Partial-Thickness Tears only).
  Participants
    Grade 1: Low (< 3 mm): number analyzed (Participants) | 33 | 0 | 33
    Grade 1: Low (< 3 mm) | 0 | 0 | 0
    Grade 2: Intermediate (3-6 mm): number analyzed (Participants) | 33 | 0 | 33
    Grade 2: Intermediate (3-6 mm) | 12 | 0 | 12
    Grade 3: High (> 6 mm): number analyzed (Participants) | 33 | 0 | 33
    Grade 3: High (> 6 mm) | 21 | 0 | 21
Tear Size: Full Thickness ONLY [Count of Participants; unit: Participants] — Full Thickness Tear Size categorized according to Cofield classification:
  * Small (less than 1 centimeter)
  * Medium (1-3 centimeters)
  * Large (3-5 centimeters)
  * Massive (greater than 5 centimeters).
  Full Thickness Tear size assessed by magnetic resonance imaging (MRI). Population: Partial-Thickness Tear not classified using this measurement (i.e. measure applies to Full Thickness Tears only).
  Participants
    Small (< 1 cm): number analyzed (Participants) | 0 | 115 | 115
    Small (< 1 cm) | 0 | 0 | 0
    Medium (1-3 cm): number analyzed (Participants) | 0 | 115 | 115
    Medium (1-3 cm) | 0 | 66 | 66
    Large (3-5 cm): number analyzed (Participants) | 0 | 115 | 115
    Large (3-5 cm) | 0 | 49 | 49
    Massive (> 5 cm): number analyzed (Participants) | 0 | 115 | 115
    Massive (> 5 cm) | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Tendon Thickness
Description: The total thickness of the tendon and any newly induced tissue at the implant site were measured at 3 months, 1 year, and 2 years using magnetic resonance imaging (MRI). Measurements were compared to pre-operative (baseline) supraspinatus tendon thickness to calculate the mean (± SD) change in post-operative supraspinatus tendon thickness by partial-thickness tear size (Intermediate or High) or full thickness tear size (Medium or Large).
Time Frame: Pre-operatively (baseline) to 3 month, 1 year, and 2 year
Population: Participants with partial-thickness or full thickness tears that provided data at the specified time frames.
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- Intermediate Partial-Thickness Tear: Intermediate partial-thickness tear (3-6 mm) of the supraspinatus tendon surgically treated by implantation of the bioinductive implant.
- High Partial-Thickness Tear: High partial-thickness tear (> 6 mm) of the supraspinatus tendon surgically treated by implantation of the bioinductive implant.
- Medium Full Thickness Tear: Medium full thickness tear (1-3 cm) of the supraspinatus tendon surgically treated by implantation of the bioinductive implant.
- Large Full Thickness Tear: Large full thickness tear (3-5 cm) of the supraspinatus tendon surgically treated by implantation of the bioinductive implant.
Arm/Group | Intermediate Partial-Thickness Tear | High Partial-Thickness Tear | Medium Full Thickness Tear | Large Full Thickness Tear
Number analyzed (Participants) | 12 | 21 | 58 | 38
millimeters
  Change from Baseline to 3 Month: number analyzed (Participants) | 12 | 21 | 53 | 37
  Change from Baseline to 3 Month | 1.7 (1.5) | 2.6 (19) | 1.2 (1.7) | 1.2 (2.2)
  Change from Baseline to 1 Year: number analyzed (Participants) | 12 | 19 | 50 | 38
  Change from Baseline to 1 Year | 1.4 (1.3) | 2.3 (1.8) | 0.6 (1.9) | 0.7 (2.2)
  Change from Baseline to 2 Year: number analyzed (Participants) | 11 | 18 | 48 | 28
  Change from Baseline to 2 Year | 1.2 (1.3) | 1.8 (2.2) | 0.7 (2.0) | 0.7 (2.3)
  Change from 3 Months to 1 Year: number analyzed (Participants) | 12 | 20 | 58 | 36
  Change from 3 Months to 1 Year | -0.3 (0.4) | -0.4 (0.6) | -0.5 (1.3) | -0.4 (1.9)
  Change from 3 Months to 2 Year: number analyzed (Participants) | 11 | 19 | 55 | 27
  Change from 3 Months to 2 Year | -0.3 (0.4) | -0.8 (1.2) | -0.6 (1.6) | -0.6 (1.8)
  Change from 1 Year to 2 Year: number analyzed (Participants) | 11 | 19 | 55 | 27
  Change from 1 Year to 2 Year | -0.1 (0.3) | -0.4 (0.9) | -0.2 (0.9) | -0.1 (1.1)

2. Primary Outcome: Integration of Induced Tissue With Underlying Tendon
Description: Partial-thickness tears were classified as Intermediate (3-6 mm) or High (> 6 mm) grade tears. Full thickness tears were categorized using Cofield classification as Medium (1-3 cm) or Large (3-5 cm). Integration and maturation of the newly induced tissue was assessed by MRI at each post-operative follow-up and determined by answering Yes, No, or Unable to determine to the following questions:
  1. Is there a visible boundary between the collagen scaffold/new tissue and the supraspinatus tendon?
  2. Is there visible evidence of a good margin between the collagen scaffold/new tissue and the deltoid?
  3. Was there evidence of bursitis in the shoulder?
  4. Does the new tissue resemble normal tendon tissue?
  5. Does the underlying tendon resemble normal tendon tissue?
  6. Is there any new defect (i.e., loss in supraspinatus tendon continuity; re-tear)?
Time Frame: 3 months, 1 year, and 2 years
Population: Participants with partial-thickness tear or full thickness tear that provided data for the specified time frames.
Measure: Count of Participants; unit: Participants
Arm/Group | Intermediate Partial-Thickness Tear | High Partial-Thickness Tear | Medium Full Thickness Tear | Large Full Thickness Tear
Number analyzed (Participants) | 12 | 21 | 66 | 48
Participants
  3 Month: Visible boundary between the collagen scaffold/new tissue and the supraspinatus tendon?: number analyzed (Participants) | 12 | 21 | 65 | 47
  3 Month: Visible boundary between the collagen scaffold/new tissue and the supraspinatus tendon?: Yes | 2 | 0 | 8 | 2
  3 Month: Visible boundary between the collagen scaffold/new tissue and the supraspinatus tendon?: No | 7 | 18 | 14 | 7
  3 Month: Visible boundary between the collagen scaffold/new tissue and the supraspinatus tendon?: Unable to determine | 3 | 3 | 43 | 38
  1 Year: Visible boundary between the collagen scaffold/new tissue and the supraspinatus tendon?: number analyzed (Participants) | 12 | 20 | 65 | 48
  1 Year: Visible boundary between the collagen scaffold/new tissue and the supraspinatus tendon?: Yes | 0 | 0 | 0 | 0
  1 Year: Visible boundary between the collagen scaffold/new tissue and the supraspinatus tendon?: No | 5 | 11 | 5 | 5
  1 Year: Visible boundary between the collagen scaffold/new tissue and the supraspinatus tendon?: Unable to determine | 7 | 9 | 60 | 43
  2 Years: Visible boundary between the collagen scaffold/new tissue and the supraspinatus tendon?: number analyzed (Participants) | 11 | 20 | 62 | 40
  2 Years: Visible boundary between the collagen scaffold/new tissue and the supraspinatus tendon?: Yes | 0 | 0 | 0 | 0
  2 Years: Visible boundary between the collagen scaffold/new tissue and the supraspinatus tendon?: No | 2 | 7 | 2 | 2
  2 Years: Visible boundary between the collagen scaffold/new tissue and the supraspinatus tendon?: Unable to determine | 9 | 13 | 60 | 38
  3 Month: Visible evidence of a good margin between the collagen scaffold/new tissue and the deltoid?: number analyzed (Participants) | 12 | 21 | 65 | 47
  3 Month: Visible evidence of a good margin between the collagen scaffold/new tissue and the deltoid?: Yes | 8 | 12 | 39 | 24
  3 Month: Visible evidence of a good margin between the collagen scaffold/new tissue and the deltoid?: No | 1 | 0 | 0 | 0
  3 Month: Visible evidence of a good margin between the collagen scaffold/new tissue and the deltoid?: Unable to determine | 3 | 9 | 26 | 23
  1 Year: Visible evidence of a good margin between the collagen scaffold/new tissue and the deltoid?: number analyzed (Participants) | 12 | 21 | 65 | 48
  1 Year: Visible evidence of a good margin between the collagen scaffold/new tissue and the deltoid?: Yes | 4 | 6 | 8 | 10
  1 Year: Visible evidence of a good margin between the collagen scaffold/new tissue and the deltoid?: No | 0 | 0 | 0 | 0
  1 Year: Visible evidence of a good margin between the collagen scaffold/new tissue and the deltoid?: Unable to determine | 8 | 15 | 57 | 38
  2 Years: Visible evidence of a good margin between the collagen scaffold/new tissue and the deltoid?: number analyzed (Participants) | 11 | 20 | 62 | 40
  2 Years: Visible evidence of a good margin between the collagen scaffold/new tissue and the deltoid?: Yes | 1 | 4 | 11 | 8
  2 Years: Visible evidence of a good margin between the collagen scaffold/new tissue and the deltoid?: No | 0 | 0 | 0 | 0
  2 Years: Visible evidence of a good margin between the collagen scaffold/new tissue and the deltoid?: Unable to determine | 10 | 16 | 51 | 32
  3 Month: Was there evidence of bursitis in the shoulder?: number analyzed (Participants) | 12 | 21 | 65 | 48
  3 Month: Was there evidence of bursitis in the shoulder?: Yes | 12 | 21 | 65 | 48
  3 Month: Was there evidence of bursitis in the shoulder?: No | 0 | 0 | 0 | 0
  3 Month: Was there evidence of bursitis in the shoulder?: Unable to determine | 0 | 0 | 0 | 0
  1 Year: Was there evidence of bursitis in the shoulder?: Yes | 12 | 21 | 66 | 48
  1 Year: Was there evidence of bursitis in the shoulder?: No | 0 | 0 | 0 | 0
  1 Year: Was there evidence of bursitis in the shoulder?: Unable to determine | 0 | 0 | 0 | 0
  2 Years: Was there evidence of bursitis in the shoulder?: number analyzed (Participants) | 11 | 20 | 62 | 40
  2 Years: Was there evidence of bursitis in the shoulder?: Yes | 10 | 18 | 57 | 40
  2 Years: Was there evidence of bursitis in the shoulder?: No | 1 | 2 | 5 | 0
  2 Years: Was there evidence of bursitis in the shoulder?: Unable to determine | 0 | 0 | 0 | 0
  3 Month: Does the new tissue resemble normal tendon tissue?: number analyzed (Participants) | 12 | 21 | 66 | 47
  3 Month: Does the new tissue resemble normal tendon tissue?: Yes | 0 | 0 | 0 | 0
  3 Month: Does the new tissue resemble normal tendon tissue?: No | 12 | 21 | 65 | 45
  3 Month: Does the new tissue resemble normal tendon tissue?: Unable to determine | 0 | 0 | 1 | 2
  1 Year: Does the new tissue resemble normal tendon tissue?: number analyzed (Participants) | 12 | 21 | 65 | 48
  1 Year: Does the new tissue resemble normal tendon tissue?: Yes | 0 | 0 | 0 | 0
  1 Year: Does the new tissue resemble normal tendon tissue?: No | 12 | 21 | 65 | 43
  1 Year: Does the new tissue resemble normal tendon tissue?: Unable to determine | 0 | 0 | 0 | 5
  2 Years: Does the new tissue resemble normal tendon tissue?: number analyzed (Participants) | 11 | 20 | 62 | 40
  2 Years: Does the new tissue resemble normal tendon tissue?: Yes | 0 | 0 | 0 | 0
  2 Years: Does the new tissue resemble normal tendon tissue?: No | 11 | 20 | 60 | 37
  2 Years: Does the new tissue resemble normal tendon tissue?: Unable to determine | 0 | 0 | 2 | 3
  3 Month: Does the underlying tendon resemble normal tendon tissue?: Yes | 0 | 0 | 0 | 0
  3 Month: Does the underlying tendon resemble normal tendon tissue?: No | 12 | 21 | 66 | 48
  3 Month: Does the underlying tendon resemble normal tendon tissue?: Unable to determine | 0 | 0 | 0 | 0
  1 Year: Does the underlying tendon resemble normal tendon tissue?: Yes | 0 | 0 | 0 | 0
  1 Year: Does the underlying tendon resemble normal tendon tissue?: No | 12 | 21 | 66 | 48
  1 Year: Does the underlying tendon resemble normal tendon tissue?: Unable to determine | 0 | 0 | 0 | 0
  2 Years: 3 Month: Does the underlying tendon resemble normal tendon tissue?: number analyzed (Participants) | 11 | 20 | 62 | 40
  2 Years: 3 Month: Does the underlying tendon resemble normal tendon tissue?: Yes | 0 | 0 | 0 | 0
  2 Years: 3 Month: Does the underlying tendon resemble normal tendon tissue?: No | 11 | 20 | 60 | 40
  2 Years: 3 Month: Does the underlying tendon resemble normal tendon tissue?: Unable to determine | 0 | 0 | 2 | 0
  3 Month: Is there any new defect (i.e., loss in supraspinatus tendon continuity; re-tear)?: Yes | 1 | 2 | 13 | 21
  3 Month: Is there any new defect (i.e., loss in supraspinatus tendon continuity; re-tear)?: No | 11 | 19 | 52 | 24
  3 Month: Is there any new defect (i.e., loss in supraspinatus tendon continuity; re-tear)?: Unable to determine | 0 | 0 | 1 | 3
  1 Year: Is there any new defect (i.e., loss in supraspinatus tendon continuity; re-tear)?: Yes | 4 | 9 | 43 | 29
  1 Year: Is there any new defect (i.e., loss in supraspinatus tendon continuity; re-tear)?: No | 8 | 9 | 20 | 19
  1 Year: Is there any new defect (i.e., loss in supraspinatus tendon continuity; re-tear)?: Unable to determine | 0 | 3 | 3 | 0
  2 Years: Is there any new defect (i.e., loss in supraspinatus tendon continuity; re-tear)?: number analyzed (Participants) | 11 | 20 | 62 | 40
  2 Years: Is there any new defect (i.e., loss in supraspinatus tendon continuity; re-tear)?: Yes | 6 | 10 | 49 | 22
  2 Years: Is there any new defect (i.e., loss in supraspinatus tendon continuity; re-tear)?: No | 4 | 8 | 13 | 18
  2 Years: Is there any new defect (i.e., loss in supraspinatus tendon continuity; re-tear)?: Unable to determine | 1 | 2 | 0 | 0

3. Primary Outcome: Fill-In of Partial Thickness Tears and Underlying Tendon Quality
Description: For tendon defects treated by standalone use of the device (i.e., implantation without surgical repair using sutures/suture anchors), post-operative follow-up MRIs will be used to estimate the amount of defect fill-in with newly induced tissue and the quality of the filled-in tissue. In the absence of fill-in with newly induced tissue, defect progression (i.e., change in size relative to previous MRIs) will be assessed. The amount of fill-in relative to the pre-operative, baseline MRI classified as:
  * 0 to <25%
  * 25% to <50%
  * 50% to < 75%
  * 75% to < 100%
  * 100%
Time Frame: 3 months, 1 year, and 2 years
Population: Only participants with partial-thickness tears that provided data for the specified time frame. Participants with Full Thickness Tears were not assessed as data for this outcome measure can only be obtained from participants with a Partial-Thickness Tear (i.e., participants with full thickness tears cannot provide fill-in partial thickness tear information needed for this outcome).
Measure: Count of Participants; unit: Participants
Arm/Group | Intermediate Partial-Thickness Tear | High Partial-Thickness Tear
Number analyzed (Participants) | 12 | 20
Participants
  3 Months: 0 to < 25% | 1 | 0
  3 Months: 25% to < 50% | 0 | 2
  3 Months: 50% to < 75% | 1 | 3
  3 Months: 75% to < 100% | 8 | 11
  3 Months: 100% | 2 | 4
  1 Year: 0 to < 25% | 0 | 1
  1 Year: 25% to < 50% | 1 | 0
  1 Year: 50% to < 75% | 2 | 3
  1 Year: 75% to < 100% | 7 | 10
  1 Year: 100% | 2 | 6
  2 Years: number analyzed (Participants) | 11 | 19
  2 Years: 0 to < 25% | 0 | 1
  2 Years: 25% to < 50% | 1 | 2
  2 Years: 50% to < 75% | 2 | 2
  2 Years: 75% to < 100% | 8 | 11
  2 Years: 100% | 0 | 3

4. Primary Outcome: Number of Participants With a Re-Tear
Description: Re-tear rate following rotator cuff repair assessed by MRI. Any new observable defect (i.e. loss in supraspinatus tendon continuity) will be classified as a re-tear.
Time Frame: 3 months, 1 year, and 2 years
Population: Participants with partial-thickness tear or full thickness tear that provided data for the specified time frames.
Measure: Count of Participants; unit: Participants
Arm/Group | Intermediate Partial-Thickness Tear | High Partial-Thickness Tear | Medium Full Thickness Tear | Large Full Thickness Tear
Number analyzed (Participants) | 12 | 21 | 66 | 49
Participants
  3 Months | 0 | 1 | 3 | 10
  1 Year | 0 | 1 | 7 | 12
  2 Years: number analyzed (Participants) | 11 | 20 | 61 | 40
  2 Years | 0 | 1 | 7 | 14

5. Secondary Outcome: Procedure Parameters: Device Implant Time
Description: Mean (± SD) device implant time in minutes was assessed starting at time from introduction of the guide wire instrument into the subacromial space through completion of the last staple.
Time Frame: Intraoperative
Population: Participants with partial-thickness tear or full thickness tear that provided data for the specified time frames.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Full Thickness Tear: Medium or large full-thickness tear (FTT) of the supraspinatus tendon surgically treated with the bioinductive implant adjunctive to surgical repair.
  Surgical repair: Surgical repair with commercially-available sutures/suture anchors.
Arm/Group | Partial-Thickness Tear | Full Thickness Tear
Number analyzed (Participants) | 33 | 115
minutes | 28.00 (16.65) | 10.50 (12.67)

6. Secondary Outcome: Procedure Parameters: Procedure Technical Success
Description: Procedure technical success was measured by the count of participants where the device was successfully delivered and affixed to the target tendon location (i.e., implant of device was attempted and successful).
Time Frame: Intraoperative
Population: Participants with partial-thickness tear or full thickness tear that provided data for the specified time frames.
Measure: Count of Participants; unit: Participants
Arm/Group | Partial-Thickness Tear | Full Thickness Tear
Number analyzed (Participants) | 33 | 115
Participants
  Device Implant Successful | 33 | 115
  Device Implant NOT Successful | 0 | 0

7. Secondary Outcome: American Shoulder and Elbow Society (ASES) Score
Description: The ASES consisted of subcomponent scores including pain, shoulder function, and shoulder scores as follows:
  1. ASES Pain Score ranges from 0 to 10, with 0 being no pain and 10 being the worst pain (lower score better).
  2. ASES Shoulder Function Score ranges from 0 to 30, with 0 being no function and 30 being full function (higher score better).
  3. ASES Shoulder Score ranges from 10 to 100, with 0 being no function and 100 being normal function (higher score better).
  Scores were collected at baseline and each successive follow-up visits (3 months, 1 year, and 2 years).
Time Frame: Baseline, 3 month, 1 year, and 2 years
Population: Participants with partial-thickness tear or full thickness tear that provided data for the specified time frames.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intermediate Partial-Thickness Tear | High Partial-Thickness Tear | Medium Full Thickness Tear | Large Full Thickness Tear
Number analyzed (Participants) | 12 | 21 | 66 | 49
score on a scale
  Baseline: ASES Pain Score | 4.6 (1.9) | 4 (2.7) | 4.8 (2.3) | 5.2 (2.6)
  3 Month: ASES Pain Score | 1.8 (1.9) | 1.3 (1.6) | 1.8 (2.2) | 1.7 (2)
  1 Year: ASES Pain Score: number analyzed (Participants) | 12 | 21 | 66 | 48
  1 Year: ASES Pain Score | 1.2 (1.6) | 0.2 (0.5) | 0.5 (1.2) | 0.5 (1.4)
  2 Years: ASES Pain Score: number analyzed (Participants) | 11 | 20 | 63 | 41
  2 Years: ASES Pain Score | 0.2 (0.4) | 0.3 (0.7) | 0.2 (0.8) | 0.5 (1.2)
  Baseline: Shoulder Function Score: number analyzed (Participants) | 12 | 20 | 66 | 46
  Baseline: Shoulder Function Score | 15.3 (5.4) | 18 (8.5) | 15.9 (5.7) | 14.2 (6.4)
  3 Month: Shoulder Function Score: number analyzed (Participants) | 11 | 17 | 66 | 45
  3 Month: Shoulder Function Score | 17 (7) | 21.1 (8) | 14.6 (6.7) | 15.6 (7.2)
  1 Year: Shoulder Function Score: number analyzed (Participants) | 11 | 17 | 64 | 47
  1 Year: Shoulder Function Score | 27 (4) | 26.8 (6.8) | 27.8 (4.2) | 27.4 (5.8)
  2 Years: Shoulder Function Score: number analyzed (Participants) | 11 | 20 | 63 | 41
  2 Years: Shoulder Function Score | 27.7 (3.4) | 26.6 (9.1) | 27.9 (6.6) | 29.2 (1.9)
  Baseline: Shoulder Score: number analyzed (Participants) | 12 | 20 | 66 | 46
  Baseline: Shoulder Score | 52.5 (13.6) | 60.9 (19.9) | 52.4 (18.3) | 48 (19)
  3 Month: Shoulder Score: number analyzed (Participants) | 12 | 17 | 66 | 45
  3 Month: Shoulder Score | 70.2 (18.6) | 78.9 (18.4) | 65.2 (19.6) | 67.9 (16.9)
  1 Year: Shoulder Score: number analyzed (Participants) | 11 | 17 | 64 | 47
  1 Year: Shoulder Score | 89.2 (14.4) | 93.7 (11.7) | 94.3 (11.6) | 93.1 (13.2)
  2 Years: Shoulder Score: number analyzed (Participants) | 11 | 20 | 63 | 41
  2 Years: Shoulder Score | 95.3 (5.8) | 92.8 (15.3) | 95.6 (13.2) | 96.3 (8.1)

8. Secondary Outcome: Constant-Murley Shoulder (CMS) Score
Description: The overall CMS shoulder score ranges from 0 to 100, with 0 being severe restrictions and 100 being no restrictions (i.e., higher score is better). Scores were collected a baseline and each subsequent follow-up (3 months, 1 year, and 2 years).
Time Frame: Baseline, 3 months, 1 year, and 2 years
Population: Participants with partial-thickness tear or full thickness tear that provided data for the specified time frames.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intermediate Partial-Thickness Tear | High Partial-Thickness Tear | Medium Full Thickness Tear | Large Full Thickness Tear
Number analyzed (Participants) | 12 | 20 | 64 | 46
score on a scale
  Baseline | 51.6 (5.6) | 58.9 (19.6) | 51.2 (16.8) | 48.5 (18.1)
  3 Months: number analyzed (Participants) | 5 | 16 | 21 | 13
  3 Months | 51.5 (13.8) | 73.7 (15.2) | 63.2 (16.8) | 65.2 (14.7)
  1 Year: number analyzed (Participants) | 10 | 18 | 61 | 46
  1 Year | 82.2 (10.4) | 85.6 (11.3) | 79.1 (11.8) | 85.3 (9.6)
  2 Years: number analyzed (Participants) | 10 | 18 | 58 | 37
  2 Years | 83.3 (9.9) | 93.8 (6) | 83.7 (9.5) | 84.4 (9.5)

9. Secondary Outcome: Recovery: Sling Time
Description: Cumulative number of days index shoulder was in a sling.
Time Frame: Post-operatively to study completion, approximately 2 years
Population: Participants with partial-thickness tear or full thickness tear that provided data for the specified time frame.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intermediate Partial-Thickness Tear | High Partial-Thickness Tear | Medium Full Thickness Tear | Large Full Thickness Tear
Number analyzed (Participants) | 12 | 21 | 64 | 49
days | 19.90 (9.39) | 26.60 (15.94) | 44.60 (43.23) | 39.20 (20.70)

10. Secondary Outcome: Recovery: Rehabilitation Time
Description: Cumulative number of completed rehabilitation or physical therapy (PT) visits in days to treat index shoulder.
Time Frame: Post-operatively to study completion, approximately 2 years
Population: Participants with partial-thickness tear or full thickness tear that provided data for the specified time frame.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intermediate Partial-Thickness Tear | High Partial-Thickness Tear | Medium Full Thickness Tear | Large Full Thickness Tear
Number analyzed (Participants) | 12 | 19 | 60 | 47
days | 14.30 (7.19) | 21.20 (11.08) | 22.50 (11.01) | 21.80 (14.44)

11. Secondary Outcome: Recovery: Return to Work
Description: Cumulative number of days between discharge and return to work (employed subjects only).
Time Frame: Post-operatively to study completion, approximately 2 years
Population: Participants with partial-thickness tear or full thickness tear that provided data for the specified time frame.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intermediate Partial-Thickness Tear | High Partial-Thickness Tear | Medium Full Thickness Tear | Large Full Thickness Tear
Number analyzed (Participants) | 12 | 21 | 44 | 36
days | 46.00 (62.99) | 58.80 (108.70) | 50.00 (72.93) | 66.50 (83.72)

12. Secondary Outcome: Recovery: Return to Normal Daily Activities
Description: Return to normal daily activities (i.e. full, unrestricted activity) determined by the cumulative number of days between discharge and return to normal daily activity.
Time Frame: Post-operatively to study completion, approximately 2 years
Population: Participants with partial-thickness tear or full thickness tear that provided data for the specified time frame.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intermediate Partial-Thickness Tear | High Partial-Thickness Tear | Medium Full Thickness Tear | Large Full Thickness Tear
Number analyzed (Participants) | 12 | 21 | 62 | 45
days | 102.40 (99.95) | 147.30 (125.30) | 130.50 (64.45) | 130.90 (84.42)

13. Secondary Outcome: Participant Satisfaction
Description: Self-reported measure of the level of satisfaction with the surgical outcome of the index surgery on 5-point Likert scale where participants were asked to indicated the best response to being satisfied with the outcome of the study procedure from one of the following:
  * Strongly Disagree
  * Disagree
  * Neither Agree or Disagree
  * Agree
  * Strongly Agree
  "Strongly Disagree" indicated the lowest level of satisfaction and "Strongly Agree" indicated the greatest level of satisfaction.
Time Frame: 3 months, 1 year, and 2 years
Population: Participants with partial-thickness tear or full thickness tear that provided data for the specified time frames.
Measure: Count of Participants; unit: Participants
Arm/Group | Intermediate Partial-Thickness Tear | High Partial-Thickness Tear | Medium Full Thickness Tear | Large Full Thickness Tear
Number analyzed (Participants) | 12 | 20 | 66 | 49
Participants
  3 Month: Strongly Disagree | 0 | 0 | 0 | 1
  3 Month: Disagree | 0 | 0 | 0 | 0
  3 Month: Neither Agree or Disagree | 2 | 3 | 4 | 2
  3 Month: Agree | 6 | 7 | 13 | 11
  3 Month: Strongly Agree | 4 | 10 | 49 | 35
  1 Year: number analyzed (Participants) | 12 | 20 | 66 | 48
  1 Year: Strongly Disagree | 0 | 0 | 1 | 2
  1 Year: Disagree | 0 | 0 | 1 | 0
  1 Year: Neither Agree or Disagree | 1 | 1 | 0 | 0
  1 Year: Agree | 2 | 3 | 7 | 6
  1 Year: Strongly Agree | 9 | 16 | 57 | 40
  2 Year: number analyzed (Participants) | 11 | 20 | 63 | 41
  2 Year: Strongly Disagree | 1 | 1 | 1 | 1
  2 Year: Disagree | 0 | 0 | 0 | 0
  2 Year: Neither Agree or Disagree | 2 | 2 | 0 | 1
  2 Year: Agree | 1 | 1 | 3 | 0
  2 Year: Strongly Agree | 7 | 16 | 59 | 39

ADVERSE EVENTS:
Time Frame: Time of enrollment (i.e. intra-operative confirmation of eligibility) through end of the study (2 year follow-up visit).
Description: Only non-serious Adverse Events (AEs) classified by the Investigator as either device-related or procedure-related were to be reported, all Serious Adverse Events (SAEs) regardless of relationship to the device, and all Unanticipated Serious Adverse Device Effects (USADEs) were to be reported per protocol. However, all Serious & Other AEs regardless of device/procedure relationship have been reported as provided. AEs were collected by investigator assessment, MRIs, and patient self-reporting.
Arm/Group | Partial-Thickness Tear | Full Thickness Tear
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/115
Serious Adverse Events (participants affected / at risk) | 1/33 | 12/115
Other Adverse Events (participants affected / at risk) | 7/33 | 10/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Partial-Thickness Tear (N=33) | Full Thickness Tear (N=115)
Cardiac Ablation (Cardiac disorders) | 1 (1) | 0 (0) — Unrelated to device and procedure
Index shoulder new rotator cuff tear and lack of healing (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Unrelated to device and procedure
Contralateral shoulder distal clavical excision, RCT debridement of degenerative labrum & bursectomy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Unrelated to device and procedure
Index shoulder recurrent rotator cuff tear (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) — Unrelated to device and procedure
Index shoulder recurrent full thickness rotator cuff tear (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Unrelated to device and procedure
Foot Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Unrelated to device and procedure
Contralateral Rotator Cuff Tear (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Unrelated to device and procedure
Index shoulder swelling and drainage (Product Issues) | 0 (0) | 1 (1) — Possibly related to device and procedure
Index shoulder pain, inflammatory changes, and osteopenia in the region of the greater tuberosity (Product Issues) | 0 (0) | 1 (1) — Possibly related to device and procedure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Partial-Thickness Tear (N=33) | Full Thickness Tear (N=115)
Midthoracic pain; slow heartbeat; R clavicle nondisplaced fracture w/fibrous union & bone formation (Cardiac disorders) | 0 (0) | 1 (1) — Unrelated to device and procedure
Index shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Unrelated to device and procedure
Index shoulder pain and stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Unrelated to device and procedure
Leg trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Unrelated to device and procedure
Contralateral shoulder ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Unrelated to device and procedure
Contralateral shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Unrelated to device and procedure
Index shoulder subacromial fluid collection/inflammation (Product Issues) | 1 (1) | 0 (0) — Possibly related to device and procedure
Index shoulder pain and stiffness (Product Issues) | 1 (1) | 0 (0) — Possibly related to device and procedure
Index shoulder bicep tendonitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Unrelated to device and possibly related to procedure
Index shoulder rash (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Unrelated to device and definitely related to procedure
Index shoulder superficial stitch abscess with continued wound drainage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Unrelated to device and definitely related to procedure
Index shoulder asymptomatic recurrent rotator cuff tear (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Unrelated to device and possibly related to procedure
Index shoulder pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Unrelated to device and definitely related to procedure
Index shoulder proximal long-head biceps rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Unrelated to device and possibly related to procedure
Index shoulder pain (Product Issues) | 0 (0) | 1 (1) — Possibly related to device and definitely related to procedure
Index shoulder recurrent rotator cuff tear (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Unrelated to device and possibly related to procedure

LIMITATIONS AND CAVEATS:
Limitations of the study include minimal source data verification, limited safety event collection due to protocol definition, the independent Sponsor safety review occurred after data was locked and extracted from the database due to acquisition integration process.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For multicenter studies the study data and results will be pooled and analyzed. If a multicenter publication is not submitted within 24 months after conclusion of study, site/investigator may publish individual results. Proposed publication must be submitted to sponsor no later than 90 prior to submission. Sponsor has right within 60 days to modify proposed publication if it will disclose patentable items.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT02200939/Prot_SAP_000.pdf